CLINICAL TRIAL: NCT03021265
Title: The Special Drug Use-results Survey on Long-term Use of Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg Fixed Dose Combination Tablets in Patients With Hypertension
Brief Title: To Evaluate Real-world Safety, Effectiveness and Appropriate Use of Micatrio® Combination Tablets Treatment in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1348.6
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T80/A5/H12.5 FDC: Patients with hypertension
  Interventions: Drug: T80/A5/H12.5 FDC

INTERVENTIONS:
Drug: T80/A5/H12.5 FDC — Drug
  Other Names: MICATRIO

SUMMARY:
Study to evaluate real-world safety, effectiveness and appropriate use of Micatrio® Combination Tablets treatment in patients with hypertension

DETAILED DESCRIPTION:
Non-interventional study based on newly collected data. The study will consist of a baseline visit and follow-up visits at Week 4, 8, 12, 24, 36 and 52 for patients who have newly initiated Micatrio® Combination Tablets. The patients will be followed up until discontinuation of Micatrio® Combination Tablets treatment or the end of study.

All patients administrated Micatrio® Combination Tablets after the launch at the sites contracted with the sponsor will be registered.

ELIGIBILITY:
Inclusion criteria:

* Patients who are prescribed with Micatrio® Combination Tablets by the discretion of investigators based on the Japanese package insert
* Patients who have never been treated with Micatrio® Combination Tablets before enrolment

Exclusion criteria:

Patients who are participating/planned to participate in a clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim; Rie Ikeda, +81364172200, Study Chair — zzCDMJP_PV_PMS@boehringer-ingelheim.com
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study based on newly collected data under real-world practice in participants with hypertension in Japan.
Pre-assignment Details: Non-randomized, post marketing surveillance, a prospective study using a continuous investigation system. No specific criteria (e.g. demographic, baseline concomitant drug in use) were defined for participant enrollment. Participants were enrolled from February 2017 to January 2018 (The first existed in Jan, system opened with delay on Feb).
Groups:
- Micatrio® Combination Tablets: Micatrio® Combination Tablets, telmisartan 80 milligram (mg)/amlodipine 5 mg/hydrochlorothiazide 12.5 mg
Period: Overall Study
Arm/Group | Micatrio® Combination Tablets
Started (Started are registered) | 676
Completed | 554
Not Completed | 122
Not completed — Adverse Event | 29
Not completed — Lack of Efficacy | 3
Not completed — Improved | 17
Not completed — Lost to Follow-up | 67
Not completed — No reason given | 2
Not completed — No visit since the first visit | 4

BASELINE CHARACTERISTICS:
Population: Safety Set: This patient set included all patients who did not have important protocol violations regarding safety and regulatory issues.
  4 patients were exclude because of missing visit after baseline
Arm/Group | Micatrio® Combination Tablets
Number analyzed (Participants) | 672
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269
  Male | 403
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Patients With Any Suspected Adverse Drug Reactions
Description: An Adverse drug reaction (ADR) is defined as an AE for which either the investigator or the sponsor (or both) assess the causal relationship to Micatrio Combination Tablets as related. The frequency of patients with any suspected ADR is presented as total number of participants with an ADR reported.
Time Frame: from first intake of Micatrio combination tablet until last intake +1 day (week 52)
Population: Safety Set: This patient set included all patients who did not have important protocol violations regarding safety and regulatory issues.
  4 patients were excluded because of missing visits after baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Micatrio® Combination Tablets
Number analyzed (Participants) | 672
Participants | 32

2. Secondary Outcome: Change From Baseline in Clinic Diastolic Blood Pressure at Week 52
Description: Change from baseline in clinic diastolic blood pressure (DBP) millimeters of mercury [mmHg] at Week 52
Time Frame: At baseline and week 52
Population: The effectiveness set included all patients in safety set with approved indication and had effectiveness information and no effectiveness related protocol violation. Only participants with data in baseline and week 52 were included in this analysis.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHG)
Arm/Group | Micatrio® Combination Tablets
Number analyzed (Participants) | 654
millimeters of mercury (mmHG) | -2.0 (10.0)

3. Secondary Outcome: Change From Baseline in Clinic Systolic Blood Pressure at Week 52
Description: Change from baseline in clinic systolic blood pressure (SBP) millimeters of mercury at Week 52
Time Frame: At baseline and week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHG)
Arm/Group | Micatrio® Combination Tablets
Number analyzed (Participants) | 654
millimeters of mercury (mmHG) | -2.6 (15.4)

ADVERSE EVENTS:
Time Frame: from first intake of Micatrio combination tablet until last intake +1 day (week 52)
Description: Safety Set: This patient set included all patients who did not have important protocol violations regarding safety and regulatory issues.
  4 patients were excluded because of missing visits after baseline.
Groups:
- Micatrio: Micatrio® Combination Tablets, telmisartan 80 milligram (mg)/amlodipine 5 mg/hydrochlorothiazide 12.5 mg
Arm/Group | Micatrio
All-Cause Mortality (participants affected / at risk) | 2/672
Serious Adverse Events (participants affected / at risk) | 20/672
Other Adverse Events (participants affected / at risk) | 0/672
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micatrio (N=672)
Gastroenteritis (Infections and infestations) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Hyperparathyroidism primary (Endocrine disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Autonomic nervous system imbalance (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Brain injury (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Blood pressure decreased (Investigations) | 1
Transcatheter aortic valve implantation (Surgical and medical procedures) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
The study was conducted in an unblinded manner and without controls. The explanatory power of the study results was limited and the study results should be interpreted with the necessary caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-10-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT03021265/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT03021265/SAP_001.pdf